CLINICAL TRIAL: NCT05725109
Title: Hepatitis C Disease Management: Diagnosis to Treatment Alerts in CHORUS™
Brief Title: Hepatitis C Diagnosis to Treatment Management
Status: Completed | Type: Observational
Sponsor: Epividian (Industry)
Collaborators: Gilead Sciences (Industry); AIDS Healthcare Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: COL2023-001
Record Dates: First submitted 2023-01-10; First posted 2023-02-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before Period (1/16/2022 to 10/17/2022): All AIDS Healthcare Foundation Healthcare Centers will be contributing to the before phase of this study. In the before phase, alerts identifying patients with active hepatitis C infection will NOT be disseminated to healthcare providers and clinic staff. Routine clinical care will be administered without knowledge of the intervention.
  Interventions: Other: Standard of Care
- After Period (1/16/2023 to 10/17/2023): All AIDS Healthcare Foundation Healthcare Centers will be contributing to the after phase of this study. In the after phase, alerts identifying patients with active hepatitis C infection will be disseminated to healthcare providers and clinic staff.
  Interventions: Other: Hepatitis C Treatment Alerts in CHORUS™

INTERVENTIONS:
Other: Hepatitis C Treatment Alerts in CHORUS™ — Clinical Health Outcomes Reporting & Utilization Service (CHORUS™) is a web-based healthcare analytics and reporting solution that transforms electronic health record data into meaningful information for healthcare providers. CHORUS™ generates a weekly email report that alerts clinics to patients with certain conditions who have a scheduled appointment in the coming week and may require close attention. CHORUS™ is a service provided to participating clinics and has been used by AIDS Healthcare Foundation for normal healthcare operations for quality improvement and retention in care in recent years. In the after period of this study, the alert will identify patients with active hepatitis C infection.
  Groups: After Period (1/16/2023 to 10/17/2023)
Other: Standard of Care — CHORUS™ is a service provided to participating clinics and has been used by AIDS Healthcare Foundation for normal healthcare operations for quality improvement and retention in care in recent years. NO alerts identifying patients with active hepatitis C infection will be disseminated.
  Groups: Before Period (1/16/2022 to 10/17/2022)

SUMMARY:
The objective of this study is to evaluate whether sending alerts to healthcare providers and clinic staff to identify patients with untreated hepatitis C infection can increase the uptake of hepatitis C treatment. A period of time without alerts will be compared to a period of time with alerts.

DETAILED DESCRIPTION:
The hepatitis C virus (HCV) is one of the most common bloodborne pathogens in the United States. A large proportion of people with HCV infection progress to chronic HCV infection despite the availability of effective treatment; chronic infection can result in cirrhosis, end-stage liver disease, liver cancer, and liver-related death. HCV infection can be cured most of the time with treatment. The objective of this before and after study is to evaluate whether sending alerts to healthcare providers and clinic staff to identify patients with untreated hepatitis C infection can increase the uptake of HCV treatment. A period of time without alerts will be compared to a period of time with alerts. Healthcare providers and clinic staff will not receive alerts during the before period of the study. Healthcare providers and clinic staff will receive alerts during the after period of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* In care at an AIDS Healthcare Foundation Healthcare Center
* Active, untreated HCV infection

Exclusion Criteria:

* <18 years of age
* Patients with active HCV infection who have a current prescription for HCV treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic Population: AIDS Healthcare Foundation Healthcare Centers across the United States and Puerto Rico are included in the study.
  Patient Population: Adult patients with active, untreated HCV infection at AIDS Healthcare Foundation Healthcare Centers are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Prescriptions for HCV treatment | End of follow-up, up to 9 months
  Proportion of patients who are prescribed HCV treatment over follow-up, out of patients with a completed visit over follow-up.

SECONDARY OUTCOMES:
HCV RNA viral load tests | End of follow-up, up to 9 months
  Frequency of HCV RNA viral load tests that occur between the first visit over follow-up and the first censoring event

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wohlfeiler, MD, Principal Investigator — AIDS Healthcare Foundation
Locations (1):
- AIDS Healthcare Foundation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No